CLINICAL TRIAL: NCT00638612
Title: AdV-tk + Valacyclovir Therapy in Combination With Surgery and Chemoradiation for Pancreas Cancer
Brief Title: AdV-tk Therapy With Surgery and Chemoradiation for Pancreas Cancer (PaTK01)
Acronym: PaTK01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Candel Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PaTK01
Record Dates: First submitted 2008-03-06; First posted 2008-03-19 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Pancreatic Adenocarcinoma; Pancreatic Cancer
Keywords: Immunotherapy; Gene Therapy; Cytotoxicity; Tumor vaccine; Radiation; Surgery; Chemoradiation
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A resectable (Experimental): Arm A is for resectable tumors. The first AdV-tk course is given prior to surgery by CT or EUS guided injection into the tumor followed by 14 days of valacyclovir. The second AdV-tk injection is into the tumor bed at the time of surgery again followed by 14 days of valacyclovir.
  Interventions: Biological: AdV-tk; Drug: Valacyclovir
- B locally advanced (Experimental): Arm B is for locally advanced tumors for which chemoradiation is the planned standard of care treatment. AdV-tk is delivered by CT or EUS guided injection into the tumor. The first AdV-tk injection is given prior to starting chemoradiation and the second in week 3 of chemoradiation. Both injections are followed by 14 days of valacyclovir.
  Enrollment has been completed for Arm B.
  Interventions: Biological: AdV-tk; Drug: Valacyclovir

INTERVENTIONS:
Biological: AdV-tk — Four dose levels of AdV-tk with a fixed dose level of valacyclovir are evaluated independently in the two arms of the study due to differences in the concomitant standard of care treatments. The first AdV-tk course is given prior to surgery or radiation by CT or EUS guided injection into the tumor followed by 14 days of valacyclovir. The second AdV-tk injection is into the tumor bed at the time of surgery in Arm A or same as the first injection in Arm B again followed by 14 days of valacyclovir. The AdV-tk dose levels are: Level 1= 3x10e10 vector particles (vp), Level 2= 1x10e11 vp, Level 3= 3x10e11 vp, Level 4= 1x10e12 vp
Drug: Valacyclovir — Valacyclovir caplets at a dose of 2 grams orally three times per day is administered for 14 days starting 1-3 days after each of the two AdV-tk injections in both arms.
  Other Names: Valtrex

SUMMARY:
The purpose of this Phase 1 study is to evaluate the safety and potential efficacy of Gene Mediated Cytotoxic Immunotherapy for pancreatic cancer. The approach uses an adenoviral vector (disabled virus) engineered to express the Herpes thymidine kinase gene (AdV-tk), followed by an antiherpetic prodrug, valacyclovir.

DETAILED DESCRIPTION:
The AdV-tk vector is injected into the tumor or tumor bed at the time of biopsy or standard tumor surgery after which valacyclovir pills are taken for 14 days. Two courses of AdV-tk, each followed by valacyclovir, are given as adjuvant to standard of care therapies (surgery and/or chemoradiation) which have been shown to work cooperatively with AdV-tk to kill tumor cells. Arm A is for resectable tumors in which the first course is given prior to surgery and the second is at the time of surgery. Arm B is for locally advanced disease in which both AdV-tk injections are administered by needle injection into the tumor before and during chemoradiation. The hypothesis is that this combination therapy can be safely delivered and will lead to improvement in the clinical outcome for patients with pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Must have presumed pancreatic adenocarcinoma based on clinical and radiologic evaluation with identifiable tumor accessible for injection (pathologic diagnosis of pancreatic adenocarcinoma must be made prior to AdV-tk injection
* For Arm A, resectable disease. Arm B for locally advanced disease has completed accrual.
* Performance status must be ECOG 0-2
* SGOT (AST)<3x upper limit of normal
* Serum creatinine<2mg/dl and calculated creatinine clearance >10ml/min
* Platelets>100,000/mm3 and WBC>3000/mm3 and ANC>1500/mm3
* Must give study specific informed consent prior to enrollment

Exclusion Criteria:

* Primary hepatic dysfunction including active hepatitis but not to exclude patients due to obstructive jaundice. If obstructive jaundice is clinically significant, bilirubin should be stable or decreasing prior to enrollment.
* Evidence of clinically significant pancreatitis as determined by the investigator.
* Patients on corticosteroids or other immunosuppressive drugs
* Known HIV+ patients
* Patients with acute infections (viral, bacterial or fungal infections requiring therapy)
* Pregnant or breast-feeding patients. Female patients of childbearing age must have negative serum or urine pregnancy test within 1 week of beginning therapy
* Evidence of distant metastatic disease at the time of enrollment or other malignancy (except squamous or basal cell skin cancers) and no prior abdominal radiation therapy or prior treatment for pancreatic cancer
* Other serious co-morbid illness or compromised organ function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-08; Primary Completion 2013-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 2 months

SECONDARY OUTCOMES:
Overall survival | 2 years
Progression free survival | 2 years
Tumor response including pathologic response | 2 months
Functional Assessment of Cancer Therapy - Pancreas (FACT-Hep) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bloomston, MD, Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - Scripps Green Hospital/Scripps Cancer Center, La Jolla, California
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aguilar LK, Shirley LA, Chung VM, Marsh CL, Walker J, Coyle W, Marx H, Bekaii-Saab T, Lesinski GB, Swanson B, Sanchez D, Manzanera AG, Aguilar-Cordova E, Bloomston M. Gene-mediated cytotoxic immunotherapy as adjuvant to surgery or chemoradiation for pancreatic adenocarcinoma. Cancer Immunol Immunother. 2015 Jun;64(6):727-36. doi: 10.1007/s00262-015-1679-3. Epub 2015 Mar 21. PMID 25795132